CLINICAL TRIAL: NCT00683904
Title: A Phase I Study of Ixabepilone in Combination With Carboplatin in Patients With Non-small Cell Lung Cancer as First-line Treatment
Brief Title: Ixabepilone in Combination With Carboplatin in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-160
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2011-04-15 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ixabepilone; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/min/mL (Active Comparator)
  Interventions: Drug: Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/min/mL
- Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/min/mL (Active Comparator)
  Interventions: Drug: Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/min/mL

INTERVENTIONS:
Drug: Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/min/mL — On Day 1 of each 21-day cycle, ixabepilone, 32 mg/m^2, intravenous (IV) solution administered as a 3-hour infusion; 30 minutes after the end of ixabepilone infusion, carboplatin, 5 mg/min/mL, intravenous IV solution infused over 30 minutes. Repeated once every 3 weeks, for a maximum of 6 cycles.
  Other Names: IXEMPRA; BMS-247550
  Arms: Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/min/mL
Drug: Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/min/mL — After all participants in Dose Level 1 (ixabepilone, 32 mg/m^2 + carboplatin, 5 mg/min/mL) have been observed for 1 full 21-day cycle, Dose Level 2(ixabepilone, 32 mg/m^2 + carboplatin, 6 mg/min/mL) opened. On Day 1 of each 21-day cycle, ixabepilone, 32 mg/m^2, IV solution administered as a 3-hour infusion; 30 minutes after the end of ixabepilone infusion, carboplatin, 6 mg/min/mL, IV solution infused over 30 minutes. Repeated once every 3 weeks, for a maximum of 6 cycles.
  Arms: Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/min/mL

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose, dose-limiting toxicity, and recommended Phase II dose of ixabepilone in combination with carboplatin in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Histologic or cytologic diagnosis of advanced non-small cell lung cancer (NSCLC)
* Advanced NSCLC, defined as stage IIIB (without indications for radiotherapy), stage IV, or recurrent
* No prior chemotherapy-containing regimens for the treatment of NSCLC
* Eastern Cooperative Oncology Group performance status of 0-1
* Life expectancy of at least 12 weeks
* Accessible for treatment and follow up; patients who could be hospitalized for first 15 days of Cycle 1
* Adequate recovery from previous systemic therapy (at least 3 weeks for surgery or radiation therapy)

Exclusion Criteria:

* Women of childbearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy for study period and for up to 4 weeks after last dose of study drug
* Women pregnant or breast feeding
* Women with a positive pregnancy test result on enrollment or prior to study drug administration
* Sexually active fertile men not using effective birth control for the entire study period and for up to 3 months after the last dose of study drug if their partners are WOCBP
* Patients with symptomatic or requiring treatment for brain metastases and/or leptomeningeal metastases
* Prior radiation must not have included ≥30% of major bone-marrow-containing areas (pelvis, lumbar spine)
* Common Terminology Criteria (CTC) Grade 2 or greater neuropathy
* Psychiatric or other disorders rendering the patient incapable of complying with protocol requirements
* Any concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix (Patients with a history of malignancy but without evidence of disease for 5 years are eligible)
* Serious uncontrolled medical disorder or active systemic infection that would impair the ability of the subject to receive protocol therapy.
* Myocardial infarction, unstable angina, or unstable congestive heart failure within 6 months
* Known history of infection with human immunodeficiency virus
* Inadequate bone marrow function
* Inadequate hepatic function
* Inadequate renal function
* Known prior severe hypersensitivity reaction (CTC Grade 2 or greater) to agents containing Cremophor®EL
* Known severe hypersensitivity reaction to agents containing carboplatin and other platinum
* Prior treatment with an epothilone and/or with platinum
* History of high-dose chemotherapy with bone marrow transplant or peripheral blood stem cell support within 2 years
* On treatment with strong Cytochrome P450 3A4 inhibitor
* Current imprisonment
* Compulsorily detention for treatment of psychiatric or physical illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-Ku, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After all participants in Dose Level 1 (ixabepilone, 32 mg/m^2 + carboplatin, 5 mg/min/mL) have been observed for 1 full 21-day cycle, Dose Level 2 (ixabepilone, 32 mg/m^2 + carboplatin, 6 mg/min/mL) opened.
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion; 30 minutes after infusion completion, carboplatin, 5 mg/min/mL, infused over 30 minutes on Day 1 of each 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL: After all participants in Dose Level 1 have been observed for 1 full 21-day cycle, Dose Level 2 opened: Ixabepilone, 32 mg/m^2, administered as a 3-hour infusion; 30 minutes after infusion completion, carboplatin, 6 mg/min/mL. infused over 30 minutes on Day 1 of each 21-day cycle.
Period: Dose Level 1
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Started | 6 | 0
Completed | 3 | 0
Not Completed | 3 | 0
Not completed — Disease progression | 2 | 0
Not completed — Adverse Event | 1 | 0
Period: Dose Level 2
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Started | 0 | 6
Completed | 0 | 4
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as a 3-hour infusion; 30 minutes after infusion completion, carboplatin, 6 mg/min/mL, infused over 30 minutes on Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (8.30) | 57.7 (10.5) | 54.4 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Japanese | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLT is defined as any of the following: Common Terminology Criteria (CTC), Version 3, Grade(Gr) 4 neutropenia (absolute neutrophil count <500 cells/mm^3) for at least 5 days or febrile neutropenia; Gr 4 thrombocytopenia (<25,000 cells/mm^3 or bleeding needing platelet transfusion); Gr 3 or 4 nausea, vomiting, or diarrhea, despite medical intervention; any other drug-related Gr 3 or 4 nonhematologic toxicity, except Gr 3 injection site reaction, fatigue/asthenia, transient arthralgia/myalgia, or transient electrolytes abnormal. Gr 1=Mild; Gr 2=Moderate; Gr 3=Severe; Gr 4=Life-threatening.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All participants who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: Participants
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion, plus carboplatin, 5 mg/min/mL, infused 30 minutes after completion of carboplatin infusion and over 30 minutes on Day 1 of each 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion, plus carboplatin, 6 mg/min/mL, infused 30 minutes after completion of carboplatin infusion and over 30 minutes on Day 1 of each 21-day cycle.
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose of Carboplatin in Combination With Ixabepilone, 32 mg/m^2
Description: The MTD was defined as the highest dose evaluated for which less than one sixth of patients experience a DLT in Cycle 1. The recommended phase 2 dose is the MTD defined in Cycle 1, with consideration given to chronic cumulative toxicity occurring at later cycles.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All participants who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: mg/min/mL
Groups:
- All Treated: All subjects who received at least 1 dose of either ixabepilone or carboplatin
Arm/Group | All Treated
Number analyzed (Participants) | 12
mg/min/mL | 6

3. Secondary Outcome: Number of Participants With Death as Outcome, Treatment-related Serious Adverse Events (SAEs), SAEs, Adverse Events (AEs), and Treatment-related AEs Leading to Discontinuation
Description: An SAE is any untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires inpatient hospitalization or prolongs existing hospitalization. An AE is any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. Treatment-related comprises certainly, probably, and possibly related and of unknown relationship to study drug.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All participants who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Death | 0 | 0
  Treatment-related SAEs | 0 | 0
  SAEs | 1 | 0
  AEs | 6 | 6
  Treatment-related AEs leading to discontinuation | 1 | 2

4. Secondary Outcome: Number of Participants With Grade 3 or Greater Treatment-related AEs
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. AEs graded according to CTC, Version 3.0. Gr 1=Mild; Gr 2=Moderate; Gr 3=Severe; Gr 4=Life-threatening. Treatment-related comprises certainly, probably, and possibly related and of unknown relationship to study drug.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All subjects who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: Participants
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin 5 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion; 30 minutes after infusion completion, carboplatin, 5 mg/min/mL, infused over 30 minutes on Day 1 of each 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Carboplatin 6 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion; 30 minutes after infusion completion, carboplatin, 6 mg/min/mL, infused over 30 minutes on Day 1 of each 21-day cycle.
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Neutropenia | 5 | 4
  Leukopenia | 4 | 4
  Anemia | 4 | 1
  Thrombocytopenia | 2 | 1
  Lymphopenia | 2 | 0
  Nausea | 0 | 1
  Liver function test abnormality | 0 | 1
  Deep vein thrombosis | 0 | 1

5. Secondary Outcome: Number of Participants With Abnormalities in Hematology Laboratory Values by Worst CTC Grade
Description: LLN=lower level of normal; ULN=upper level of normal. Hemoglobin (g/dL; LLN=11.3; ULN=14.9); leukocytes (*10^3 c/uL; LLN=4.1; ULN=6.1); lymphocytes (*10^3 c/uL); neutrophils (absolute), neutrophils + bands (*10^3 c/uL); platelet count (*10^9 c/L; LLN=131; ULN=365)
  Appendix 7.1.2
Time Frame: At screening and Days 8 and 15 of Cycle 1 (21 days)
Population: All participants who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: Participants
Groups:
- Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion; 30 minutes after infusion completion, carboplatin, 6 mg/min/mL, infused over 30 minutes on Day 1 of each 21-day cycle.
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Hemoglobin: Grade 1 (10.0- LLN) | 0 | 0
  Hemoglobin: Grade 2 (8.0-<10.0) | 2 | 5
  Hemoglobin: Grade 3 (6.5-<8.0) | 4 | 1
  Hemoglobin: Grade 4 (<6.5) | 0 | 0
  Hemoglobin: Not reported | 0 | 0
  Leukocytes: Grade 1 (3.0-<LLN) | 0 | 0
  Leukocytes: Grade 2 (2.0-<3.0) | 2 | 1
  Leukocytes: Grade 3 (1.0-<2.0) | 4 | 5
  Leukocytes: Grade 4 (<1.0) | 0 | 0
  Leukocytes: Not reported | 0 | 0
  Lymphocytes (absolute): Grade 1 (0.8-<1.5) | 4 | 1
  Lymphocytes (absolute): Grade 2 (0.5-<0.8) | 0 | 5
  Lymphocytes (absolute): Grade 3 (0.2-<0.5) | 2 | 0
  Lymphocytes (absolute): Grade 4 (<0.2) | 0 | 0
  Lymphocytes: Not reported | 0 | 0
  Neutrophils (absolute): Grade 1 (1.5-<2.0) | 0 | 1
  Neutrophils (absolute): Grade 2 (1.0-<1.5) | 1 | 0
  Neutrophils (absolute): Grade 3 (0.5-<1.0) | 1 | 0
  Neutrophils (absolute): Grade 4 (<0.5) | 4 | 5
  Neutrophils (absolute): Not reported | 0 | 0
  Neutrophils+bands (absolute): Grade 1 (1.5-<2.0) | 0 | 1
  Neutrophils+bands (absolute): Grade 2 (1.0-<1.5) | 1 | 0
  Neutrophils+bands (absolute): Grade 3 (0.5-<1.0) | 2 | 1
  Neutrophils+bands (absolute): Grade 4 (<0.5) | 3 | 4
  Neutrophils+bands (absolute): Not reported | 0 | 0
  Platelet count: Grade 1 (75.0-<LLN) | 1 | 3
  Platelet count: Grade 2 (50.0-<75.0) | 3 | 2
  Platelet count: Grade 3 (25.0-<50.0) | 2 | 1
  Platelet count: Grade 4 (<25.0) | 0 | 0
  Platelet count: Not reported | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in Serum Chemistry Laboratory Values by Worst CTC Grade
Description: ULN=upper limit of normal; LLN=lower limit of normal. Alkaline phosphatase=ALP(LLN=115; ULN=359) (U/L); alanine aminotransferase=ALT (LLN=8; ULN=42)(U/L); aspartate aminotransferase=AST (LLN=13; ULN=33) (U/L); albumin (LLN=3.7; ULN=5.2)(g/dL); bilirubin (LLN=0.3; ULN=1.2)(mg/dL); calcium (LLN=8.7; ULN=10.3)(mg/dL); creatinine (LLN=0.6; ULN=1.1)(mg/dL); potassium (LLN=3.6; ULN=4.9) (mEq/L); sodium (LLN=138; ULN=146) (mEq/L)
Time Frame: At screening and Days 8 and 15 of Cycle 1 (21 days)
Population: All participants who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  ALT: Grade 1 ( >1.0-2.5*ULN) | 3 | 2
  ALT: Grade 2 (>2.5-5.0*ULN) | 2 | 1
  ALT: Grade 3 ( >5.0-20.0*ULN ) | 0 | 1
  Albumin: Grade 1 (<LLN-3.0) | 4 | 4
  ALP: Grade 1 ( >1.0-2.5*ULN) | 0 | 4
  AST: Grade 1 ( >1.0-2.5*ULN) | 4 | 3
  AST: Grade 2 (>2.5-5.0*ULN) | 1 | 1
  Bilirubin: Grade 1 (>1.0-1.5*ULN) | 1 | 1
  Bilirubin: Grade 2 (>1.5-3.0*ULN) | 1 | 0
  Calcium: Grade 1 (8.0-<LLN or >ULN -11.5) | 5 | 4
  Creatinine: Grade 1 (>1.0-1.5*ULN) | 0 | 2
  Potassium: Grade 1 (3.0-<LLN or >ULN-5.5) | 3 | 1
  Sodium: Grade 1 (130-<LLN or >ULN-150) | 4 | 5

7. Secondary Outcome: Number of Participants With Abnormalities in Urine Testing Results by Worst CTC Grade
Description: Toxicities graded according to CTC, Version 3. Protein Gr 1: <1.0 g/24 hrs (1+); Gr 2: 1.0 to 3.4 g/24 hrs (2+ to 3+ ); Gr 3: >=3.5 g/24 hrs (4+); Gr 4: Nephrotic syndrome. Note: + = qualitative measure of urine chemistry.
Time Frame: At screening and Days 8 and 15 of Cycle 1 (21 days)
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Protein (Grade 1) | 2 | 2
  Protein (Grade 2) | 3 | 0
  Protein (Grade 3) | 0 | 0
  Protein (Grade 4) | 0 | 0
  Not reported | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormalities in Blood Pressure and Heart Rate
Description: Blood pressure and heart rate obtained before ixabepilone infusion, every 1 hour during and at the end of ixabepilone infusion, and at the end of carboplatin infusion in Cycle 1. For subsequent cycles, vital signs obtained before ixabepilone infusion, at the end of ixabepilone infusion, and at the end of carboplatin infusion. Any new or worsening clinically significant changes since last entry were recorded as appropriate AE or SAE.
Time Frame: At screening and Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (Study day 22)
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Blood pressure | 0 | 0
  Heart rate | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormalities in Weight and Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Participants weighed same day as serum chemistry tests. Body surface area recalculated only if body weight changes >10%. ECOG criteria used to assess disease progression and affects on daily living abilities and to determine appropriate treatment and prognosis. Grade 1=Restricted physical activity but ambulatory and capable of light work; Grade 2=Ambulatory, capable of self care, but unable to carry out any work activities; Grade 3=Capable of limited self care, confined to bed or chair 50% or more of waking hours; Grade 4=Completely disabled, totally confined to bed or chair.
Time Frame: At screening of Cycle 1 (21 days) and Day 1 of Cycle 2 (Study day 22)
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Participants
  Blood pressure | 0 | 0
  Heart rate | 0 | 0
  Weight | 0 | 0
  ECOG performance status | 0 | 0

10. Secondary Outcome: Number of Participants at Each Response Evaluation Criteria in Solid Tumors (RECIST) Assessment
Description: Tumor response was assessed using the RECIST assessment: Complete response (CR)=Disappearance of all clinical and radiologic evidence of target lesions; Partial response (PR)=At least 30% reduction in the sum of the longest diameters of all target lesions; Progressive disease (PD)=At least 20% increase in the sum of the longest diameters of all target lesions; Stable disease (SD)=Neither PR nor PD criteria were met.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All treated participants with measurable disease at baseline, as determined by investigator
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 4 | 6
Participants
  CR | 0 | 0
  PR | 2 | 1
  PD | 2 | 0
  SD | 0 | 4
  Unable to be assessed (patient discontinuation) | 0 | 1

11. Secondary Outcome: Maximum Observed Plasma Concentration of Ixabepilone
Time Frame: Days 1 to 8 of Cycle 1 (21 days)
Population: All participants who received ixabepilone and carboplatin and had adequate pharmacokinetic concentration profiles
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
ng/mL | 195.77 (45.89) | 250.32 (76.17)

12. Secondary Outcome: Time of Maximum Observed Plasma Concentration of Ixabepilone
Time Frame: Days 1 to 8 of Cycle 1 (21 days)
Population: All participants who received ixabepilone and carboplatin and had adequate pharmacokinetic concentration profiles
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Hours | 2.61 (0.88) | 2.43 (1.03)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero Extrapolated to Infinite Time of Ixabepilone
Time Frame: Days 1 to 8 of Cycle 1 (21 days)
Population: All participants who received ixabepilone and carboplatin and had adequate pharmacokinetic concentration profiles
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
ng*h/mL | 1542.11 (585.29) | 2135.93 (1246.08)

14. Secondary Outcome: Volume of Distribution at Steady State of Ixabepilone
Time Frame: Days 1 to 8 of Cycle 1 (21 days)
Population: All participants who received ixabepilone and carboplatin and had adequate pharmacokinetic concentration profiles
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Liters | 1131.02 (373) | 1122.82 (477)

15. Secondary Outcome: Total Body Clearance of Ixabepilone
Time Frame: Days 1 to 8 of Cycle 1 (21 days)
Population: All participants who received ixabepilone and carboplatin and had adequate pharmacokinetic concentration profiles
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Ixabepilone, 32 mg/m^2 + Carboplatin, 5 mg/Min/mL | Ixabepilone, 32 mg/m^2 + Carboplatin, 6 mg/Min/mL
Number analyzed (Participants) | 6 | 6
Liters/hour | 33.64 (11) | 25.20 (8)

ADVERSE EVENTS:
Groups:
- Ixabepilone, 32 mg/m2 + Carboplatin 5 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion, plus carboplatin, 5 mg/min/mL, infused 30 minutes after completion of carboplatin infusion and over 30 minutes on Day 1 of each 21-day cycle.
- Ixabepilone, 32 mg/m2 + Carboplatin 6 mg/Min/mL: Ixabepilone, 32 mg/m^2, administered as 3-hour infusion, plus carboplatin, 6 mg/min/mL, infused 30 minutes after completion of carboplatin infusion and over 30 minutes on Day 1 of each 21-day cycle.
Arm/Group | Ixabepilone, 32 mg/m2 + Carboplatin 5 mg/Min/mL | Ixabepilone, 32 mg/m2 + Carboplatin 6 mg/Min/mL
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m2 + Carboplatin 5 mg/Min/mL (N=6) | Ixabepilone, 32 mg/m2 + Carboplatin 6 mg/Min/mL (N=6)
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m2 + Carboplatin 5 mg/Min/mL (N=6) | Ixabepilone, 32 mg/m2 + Carboplatin 6 mg/Min/mL (N=6)
Asthenopia (Eye disorders) | 0 | 1
Protein urine (Investigations) | 5 | 1
Weight decreased (Investigations) | 1 | 3
Blood urine present (Investigations) | 3 | 3
Glucose urine present (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 3
Blood sodium increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 2 | 1
Protein total decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 1
Blood potassium increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 4
Dysarthria (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Leukopenia (Blood and lymphatic system disorders) | 6 | 6
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 4
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Injection site reaction (General disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.